CLINICAL TRIAL: NCT05094453
Title: Borescope Visually Assisted Intubation Through Fekry Intubating Airway; a Prospective Randomized Controlled Study
Brief Title: Borescope Visually Assisted Intubation Through Fekry Intubating Airway
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Yahia El Sayed Kamel, Assistant lecturer of Anesthesia, ICU and pain management, Cairo University
Other Study IDs: Airway management
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Intubation; Difficult or Failed
Keywords: visually assisted intubation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to introduce the borescope visually assisted through Fekry oral Intubating airway as a new means of intubation.

DETAILED DESCRIPTION:
Endotracheal intubation is one of the fundamental skills that should be mastered by the anesthesiologist. One of the important causes of anesthesia related mortality and morbidity is difficult airway related events.

A key step in endotracheal intubation is the alignment of the oral, pharyngeal and laryngeal axes. More recently a 2-curve concept has been proposed, involving a primary (oro-pharyngeal curve) and a secondary (pharyngo-glotto-tracheal) curve. The need to align the visual axis to these axes is a common reason for poor visualization of the glottis and the difficulty encountered during endotracheal intubation. Video laryngoscopes (VLS) overcome this problem by allowing the viewer to see the glottis through a camera attached to a curved blade.

Several video laryngoscopes (VLS) are available in the market to facilitate endotracheal intubation. These devices are precluded by their cost and availability especially in developing countries.

Borescope is an instrument that is used to see through a small hole. The endoscope camera diameter is 5.5 mm and the cable is 1 m long with flexible fiber which could be bended as needed. It is illuminated by circumferentially arranged 6 LED lamps on the head of camera. The other end of cable is connected to Android smart phone (Samsung galaxy S5) which supports OTG (on-the-go) function.

Universal Serial Bus (USB) borescopes are commonly used in dental procedures as a dental imaging system.

Borescopes are rugged, waterproof and work on trickle power from USB ports of a laptop, computer or a Smartphone.

The Smartphone provides the power supply and processes the image. The resultant image can be viewed and recorded in any Smartphone by using a variety of free video capture available applications. The auto detect feature of Smartphones allows the image to appear as soon as the USB device is connected, thus requiring minimal time to set up. As the device is waterproof it can be easily sterilized by soap water and glutaraldehyde.

A low-cost VLS ("v-scope") using a straight Miller blade has been tried. The investigators attached an USB borescope to a Miller's blade by waterproof tapes and connected it to a smart phone via an USB-OTG (On the go) cable. Interestingly, it was compared with a conventional Miller blade for intubation and concluded that an ordinary borescope can be used as an effective VLS which is cost effective, easy to assemble and use and can provide acceptable glottis views even in the hands of non-experts.

A similar scope was described, but using a Macintosh blade, in February 2016. The device used the video processing capabilities of a personal computer to display real processing present in the ubiquitous smart phone, keeping the initial and recurring costs of the technique low.

Since economic consideration is very crucial in developing countries, this study is going to test a safe, low cost technique of visually assisted intubation using the Borescope and Fekry airway instead of the high cost offered by different video laryngoscopes (VLS) available in the market.

Fekry airway (Oral Intubating Airway; Egyptian Patent 28118):

Several modifications and versions of oro-pharyngeal airways were introduced into the market to facilitate fiberoptic intubation and easy removal of the airway after placement of ETT.

Fekry airway is a modification of the Williams airway. The modification made to the Williams airway is that the roof of the proximal cylindrical tunnel is removed thus the airway became open anteriorly. This modification offers the following advantages: it allows easy one step insertion of the tube. Also it facilitates the airway removal after ETT insertion without need to remove the international connection of the ETT. Thus Fekry airway can be easily removed from around the tube while it is connected to anesthesia machine (this reduces the risk of inadvertent ETT dislodgement during airway removal).

This study is introducing a novel way to replace the high cost videolaryngoscopy to be used for safe educational purposes and management of difficult airway scenarios.

Our hypothesis is that the borescope in association with Fekry oral airway will introduce a new means for low cost, efficient video assisted endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia residents in the last year of residency.
* Anesthesia assistant lecturers in the first year of work.

Exclusion Criteria:

* Assistant lecturers who are in the career for more than one year.
* Paramedical personnels.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll 35 anesthesia residents in their last year of residency and assistant lecturers in their first year of work who will try to intubate a manikin using the borescope visually assisted through Fekry oral Intubating airway.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the success rate of intubation | 1 June 2020 to 1 March 2021
  To evaluate the success rate of intubation using borescope visually assisted through Fekry airway.

SECONDARY OUTCOMES:
Number of intubation attempts. | 1 June 2020 to 1 March 2021
  Total number of attempts.
Total intubation time | 1 June 2020 to 1 March 2021
  starting from introduction of the borescope/ETT assembly till introducing the tube into the vocal cords reaching the carina
Need of external manipulations to visualize the view. | 1 June 2020 to 1 March 2021
  such as crcoid pressure or laryngeal manipulations

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Asswa, Professor, Study Director — Cairo University; Maha Youssef, A.Professor, Study Director — Cairo University; Inas Ali, lecturer, Study Director — Cairo University; Sahar Kassem, lecturer, Study Director — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, الجيزة, Egypt

IPD SHARING:
Plan to Share IPD: No